CLINICAL TRIAL: NCT04115891
Title: Can Lavender Oil Inhalation Help to Overcome Dental Anxiety and Pain in Children? A Randomized Clinical Trial
Brief Title: Lavender Oil Inhalation Help to Overcome Dental Anxiety Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazife Begüm KARAN, Assistant Professor, DDS, PhD, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Dental Anxiety; Anxiety Disorder; Aromatherapy
Keywords: lavandula; phytotherapy; aromatherapy; dental anxiety; anaesthesia
MeSH Terms: conditions — Anxiety Disorders | interventions — Inhalation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender oil group (Experimental): 100 % pure, high strength lavender oil inhalation in a separate room for 3 minutes, prior to tooth extractions.
  Anxiety scale (FIS) Pain scale 1 (FLACC) Pain scale 2 (WBS) Vital signs 1 (systolic and diastolic blood pressure) Vital signs 2 (heart rate) Vital signs 3 (saturation)
  Interventions: Other: Anxiety scale; Other: Pain scale - 1; Other: Pain scale - 2; Behavioral: Inhalation
- Control group (Sham Comparator): No application prior to interventions. No lavender oil inhalation.
  Anxiety scale (FIS) Pain scale 1 (FLACC) Pain scale (WBS) Vital signs 1 (systolic and diastolic blood pressure) Vital signs 2 (heart rate) Vital signs 3 (saturation)
  Interventions: Other: Anxiety scale; Other: Pain scale - 1; Other: Pain scale - 2

INTERVENTIONS:
Other: Anxiety scale — Anxiety Face Image Scale (FIS) assessment in a separate room with face to face interview.
Other: Pain scale - 1 — Face, Legs, Activity, Cry, Consolability (FLACC), to assess objective operational pain after anesthesia injection and tooth extraction
Other: Pain scale - 2 — Wong Baker Pain Rating scale (WBS), to assess subjective operational pain after anesthesia injection and tooth extraction
Behavioral: Inhalation — lavender oil inhalation in a separate room for 3 minutes prior to interventions
  Other Names: 100 % pure, high strength lavender oil inhalation
  Arms: Lavender oil group

SUMMARY:
The purpose of this study is to investigate the impact of lavender oil (Lavandula angustifolia) on anxiety, pain and vital signs (blood pressure, heart rate and saturation) among children planned to undergone surgical intervention.

DETAILED DESCRIPTION:
Lavender oil has sedative properties. Dental anxiety is one of the most common obstacles to dental care, especially for children ranges from 3% to 43% in different populations. To the best of our knowledge, this is the first study to investigate the use of lavender oil inhalation and to assess the correlation of anxiety and vital signs among children during a stressful surgical dental intervention. This study design was constructed according to the vital sign evaluations, anxiety and pain scores. Primary hypothesis was that of lavender oil inhalation prior to surgical dental interventions would affect vital signs and consequently reduce anxiety and perception of pain in children.

ELIGIBILITY:
Inclusion Criteria:

* being between 6 and 12 years of age
* children who are determined as Frankl 2, 3 or 4
* intellectually sufficient to complete the anxiety scale
* volunteer to take part in the study
* whose parents were willing to participate into the study

Exclusion Criteria:

* aged under 6
* has cognitive, cooperation (i.ex. Frankl 1) or systemic problems
* common allergies or dental pain

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Vital Sign Measurements - 1 (sistolic and diastolic blood pressure) | through study completion an average of 9 months
  changes in systolic and diastolic blood pressure pre-operatively, intra-operatively, post-operatively
Vital Sign Measurements - 2 (heart rate) | through study completion an average of 9 months
  changes in heart rate pre-operatively, intra-operatively, post-operatively
Vital Sign Measurements - 3 (saturation) | through study completion an average of 9 months
  changes in saturation pre-operatively, intra-operatively, post-operatively

SECONDARY OUTCOMES:
Anxiety Scale - Face Image Scale (FIS) | through study completion an average of 9 months
  Five cartoon faces symbolized different emotions from very happy to very unhappy. The children chose one face at which they feel most like at that moment. One point is given to most positive face and 5 point is given to most negative face.
Pain Scale 1 - Face, Legs, Activity, Cry, Consolability (FLACC) | through study completion an average of 9 months
  FLACC has five categories of behavior to rate pain as follows; facial expression, leg movement, activity, cry and consolability. The scores of each category are between 0 and 2. The total scores can change from 0 to 10 defined as mild (1-3), moderate (4-6) and severe (7-10).
Pain Scale 2 - Wong Baker Pain Rating Scales (WBS) | through study completion an average of 9 months
  WBS combines pictures and numbers to rate pain. The scale has six faces assigned numerical ratings from 0 'no hurt' to 10 'hurts worst'. Administration of WBS is easy, not time consuming and requires minimal instructions

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Nazife Begüm KARAN, Ankara, Merkez
  - Nazife Begüm KARAN, Rize, Merkez

IPD SHARING:
Plan to Share IPD: Undecided
Beginning 3 months and ending 5 years following article publication all data will be shared with other researchers